CLINICAL TRIAL: NCT06879340
Title: A Phase 1 Multicenter, Open Label Trial Evaluating the Safety and Efficacy of DuoCAR20.19.22-D95 in Adult Patients With Relapsed or Refractory B-cell Malignancies
Brief Title: Evaluating the Safety and Efficacy of DuoCAR20.19.22-D95 in Adult Patients With Relapsed or Refractory B-cell Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Joseph McGuirk, Division Director Hematologic Malignancies and Cellular Therapeutics, University of Kansas Medical Center
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00161006
Record Dates: First submitted 2025-03-03; First posted 2025-03-17 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; B-cell Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Lymphoma, B-Cell; Burkitt Lymphoma | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Phase 1 (Dose Escalation) (Experimental): Lymphodepletion:
  Fludarabine: Days -6 to -3 (4 days total) Cyclophosphamide: Days -4 and -3 (2 days total)
  Investigational Treatment:
  DuoCAR20.19.22-D95 will be infused on day # 0
  Patients will receive lymphodepletion chemotherapy and receive the CAR T cell infusion on day 0 (or up to day +14 in extenuating clinical conditions). Patients will be hospitalized inpatient period of at least 7 days from the day of the CAR T infusion.
  Interventions: Drug: DuoCAR20.19.22-D95; Drug: Fludarabine (Conditional therapy); Drug: Cyclophosphamide (Conditional therapy)

INTERVENTIONS:
Drug: DuoCAR20.19.22-D95 — Patient derived autologous T cells, lentiviral transduced to generate, using the Miltenyi CliniMACS Prodigy® closed transduction system, a Duo-CAR-T cells targeting cell surface antigens CD19/20/22.
Drug: Fludarabine (Conditional therapy) — Lymphodepletion chemotherapy
Drug: Cyclophosphamide (Conditional therapy) — Lymphodepletion chemotherapy

SUMMARY:
This multicenter phase 1 trial with "3 + 3" dose escalation design seeks to examine the feasibility and safety of the administration of autologous T cells that have been modified through the introduction of chimeric antigen receptors targeting the B cell surface antigens CD19/20/22 following administration of a chemotherapy lymphodepletion regimen in adults with relapsed/refractory B-cell acute lymphoblastic leukemia (ALL) or Non-Hodgkin's lymphoma (NHL). The overall goals of this study are to estimate maximum tolerated dose (MTD) level, establish the overall safety profile and evaluate initial efficacy of administering duo-CAR-T cell treatment in this patient population.

DETAILED DESCRIPTION:
Dose Escalation Cohort (Phase 1)

This will have 3 enrollment groups:

Group A: Participants with B-ALL (CAR pre-treated or CAR naïve), Group B: Participants with B-NHL (CAR pre-treated), Group C: Participants with B-NHL (CAR naïve)

The trial will begin with a phase I dose escalation evaluation in each of the three enrollment groups. Participants will be treated either at dose level 1 and dose level -1 or at dose level 1 and dose level 2 of CAR T cells. This phase will determine the MTD and /or RP2D for the subsequent Phase 2 study. The trial duration for an individual participant is 15 years from DUOCAR20.19.22-D95-CAR T cell infusion. Following infusion, DLT assessments will continue through end of Day 30 visit during Dose Escalation Phase 1. Efficacy and routine safety monitoring for Phase 1 cohort will occur at established protocol-defined intervals through Year 2 or until the start of a new treatment regimen, whichever occurs sooner. The observational long-term follow-up portion of the study will then become operative.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of participant to understand this study, and participant willingness to sign a written informed consent
2. Women of childbearing potential must have a negative serum pregnancy test 48 hours prior to the start of preparatory regimen
3. Patients must have histologically confirmed aggressive B-Cell NHL or ALL as stated below:

   A. Patients with relapsed or refractory B-Cell ALL i. Demonstration of one or more antigens of interest (CD19, CD20, CD22) in most recent disease evaluation prior to study entry and within 30 days of study entry.

   ii. Patients with relapsed/refractory disease in blood, marrow, and extramedullary sites including CSF will be eligible when there is immunophenotypic evidence of CD19 and/or CD20 and/or CD22 expression

   iii. Primary refractory disease at study entry defined as: A morphologic complete response has never been achieved prior to study entry.

   iv. Early first relapse at study entry defined as: Disease recurrence by morphologic assessment after duration of first remission at ≤ 18 months

   v. Relapsed Refractory disease (first or later relapse) at study entry defined as: Morphologic complete response was not achieved after initiation of a second-line (or later) systemic therapy

   vi. Second or greater relapse at study entry defined as: Any disease recurrence following a second or later complete response (with treatment history including two or more lines of systemic therapy)

   vii. Additional considerations beyond above criteria:
   * Patients with relapsed or refractory disease after allogeneic stem cell transplantation must be >100 days from HSCT to be eligible for study participation. Furthermore, post-HSCT immunosuppressive medications must be discontinued for at least 4 weeks prior to study entry
   * Prior CAR-T therapy is permissible if ≥ 3 months from therapy completion
   * Morphological disease in the bone marrow Note: Morphologic disease is defined as blasts being at least 5% in the bone marrow.

   B. Histologically confirmed aggressive B cell NHL, including the following types defined by WHO 2008 after 2 or more lines of prior therapy:

   i. DLBCL not otherwise specified; T cell/histiocyte rich large B cell lymphoma; DLBCL associated with chronic inflammation; Epstein-Barr virus (EBV)+ DLBCL of the elderly; Primary cutaneous DLBCL, leg type; OR ii. Primary mediastinal (thymic) large B cell lymphoma iii. Follicular lymphoma 3b and transformation of follicular lymphoma to DLBCL will also be included iv. High-grade B cell lymphoma v. Chemotherapy-refractory disease, defined as one or more of the following:
   * Refractory disease is defined as progressive or stable disease as the best response to the most recent prior therapy or relapse within 12 months of autologous stem cell transplantation. Two prior lines of therapy are required for LBCL eligibility. The second line therapy may be chemotherapy based, autologous stem cell transplantation, or CAR-T.
   * Relapsed or refractory disease after allogeneic transplant provided patient is at least 100 days from stem cell transplant at the time of enrollment and off of immunosuppressive medications for at least 4 weeks prior to enrollment
   * Patients must have received 2 or more lines of adequate prior therapy including at a minimum:

     * anti-CD20 monoclonal antibody unless investigator determines that tumor is CD20- negative and
     * an anthracycline containing chemotherapy regimen
     * for patients with transformed FL must have received prior chemotherapy for follicular lymphoma and subsequently have chemorefractory disease after transformation to DLBCL vi. Prior CAR T therapy permissible if ≥ 3 months from the therapy vii. At least 1 measurable lesion according to the revised IWG Response Criteria for Malignant Lymphoma (Cheson 2007). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy C. Relapsed or refractory indolent non-Hodgkin lymphoma i. Histologically confirmed indolent non-Hodgkin lymphoma, including grade 1-3b follicular lymphoma or nodal or extranodal marginal zone lymphoma (both per WHO 2016 classification criteria) ii. Relapsed or refractory disease (per Lugano criteria) after two or more previous lines of therapy, iii. Previous lines of therapy to include an anti-CD20 monoclonal antibody combined with an alkylating agent iv. Prior CAR T therapy permissible if ≥ 3 months from the therapy v. At least 1 measurable lesion according to the revised IWG Response Criteria for Malignant Lymphoma (Cheson 2007). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy vi. Relapsed or refractory disease after allogeneic transplant provided patient is at least 100 days from stem cell transplant at the time of enrollment and off of immunosuppressive medications for at least 4 weeks prior to enrollment D. Relapsed or Refractory Mantle-Cell Lymphoma i. Histologically confirmed mantle-cell lymphoma with either cyclin D1 overexpression or presence of the translocation (T11:14) ii. Disease that is either relapsed or refractory to at least 2 prior lines of previous regimens for mantle-cell lymphoma iii. Previous therapy must have included anthracycline- or bendamustine-containing chemotherapy, an anti-CD20 monoclonal antibody, and BTK inhibitor therapy
4. Prior CAR T therapy permissible if ≥ 3 months from the therapy
5. At least 1 measurable lesion according to the revised IWG Response Criteria for Malignant Lymphoma (Cheson 2007). Lesions that have been previously irradiated will be considered measurable only if progression has been documented following completion of radiation therapy
6. Relapsed or refractory disease after allogeneic transplant provided patient is ≥ 3 months from stem cell transplant at the time of enrollment and off of immunosuppressive medications for at least 4 weeks prior to enrollment
7. Meet institutional criteria for leukapheresis procedure or have availability of previously- collected and stored leukapheresis product that satisfies minimum requirements
8. Eastern cooperative oncology group (ECOG) performance status of 0 to 2.
9. Adequate hematologic and organ function NOTE: Patients with established diagnosis of benign neutropenia are eligible to participate with ANC between 1000-1500 if in the opinion of treating physician the trial treatment does not pose excessive risk of infection to the patient.
10. Adults ≥ 18 years of age, with no upper limit of age
11. Life expectancy >2 months
12. ≥ 3 months from prior CAR
13. Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence or to use the forms of contraception listed in Child-Bearing Potential/Pregnancy section from the time of signing informed consent to at least 12 months following DuoCAR20.19.22-D95 infusion and until CAR positive viable T cells are no longer present by quantitative polymerase chain reaction (qPCR) on two consecutive tests. Men must agree not to donate sperm for the same time period.

Exclusion Criteria:

1. Patients with CLL, Richter's transformation, and Burkitt lymphoma
2. Active CNS involvement by malignancy - CNS3 disease, i.e., patients with WBC count in CSF ≥5 and having blasts in the CSF in patients with ALL or detection of NHL on CSF by flow cytometry or active CNS involvement on imaging)
3. Chemotherapy other than lymphodepleting chemotherapy within 2 weeks of infusion
4. Investigational medicinal product within the last 30 days prior to screening Note: Investigational therapies must not be used at any time while on study until the first progression following DuoCAR20.19.22-D95 CAR T infusion.
5. The following medications are excluded:

   1. Steroids: Therapeutic doses of steroids must be stopped > 72 hours prior to leukapheresis and > 72 hours prior to DuoCAR20.19.22-D95 infusion. However, the following physiological replacement doses of steroids are allowed: <12 mg/m2/day hydrocortisone or equivalent
   2. Immunosuppression: Any other immunosuppressive medication must be stopped ≥ 2 weeks prior to leukapheresis and ≥ 2 weeks prior to DuoCAR20.19.22-D95 infusion. This could include check point inhibitors (monoclonal antibodies and small molecule modulators).
   3. Antiproliferative therapies other than lymphodepleting chemotherapy within 2 weeks prior to infusion
   4. Short acting drugs used to treat leukemia or lymphoma (e.g., tyrosine kinase inhibitors, and hydroxyurea) must be stopped > 72 hour prior to leukapheresis and > 72 hours prior to DuoCAR20.19.22-D95 infusion
   5. Other cytotoxic drugs, including low dose daily or weekly maintenance chemotherapy, must not be given within 2 weeks prior to leukapheresis and within 2 weeks prior to DuoCAR20.19.22-D95 infusion.
   6. Antibody use including anti-CD20 therapy within 4 weeks prior to infusion or 5 half-lives of the respective antibody, whichever is longer. Note: Rituximab is excluded within 4 weeks prior to infusion.
   7. CNS disease prophylaxis or treatment must be stopped > 1 week prior to DuoCAR20.19.22-D95 infusion (e.g., intrathecal methotrexate)
6. Prior radiation therapy within 2 weeks of infusion
7. Active replication of or prior infection with hepatitis B or active hepatitis C (HCV RNA positive)
8. HIV positive patients (excluding false positive HIV test resulting from the viral vector used in prior CAR T)
9. Uncontrolled acute life threatening bacterial, viral or fungal infection (e.g., blood culture positive ≤ 72 hours prior to infusion)
10. Unstable angina and/or myocardial infarction within 6 months prior to screening
11. Previous or concurrent malignancy with the following exceptions:

    1. Adequately treated basal cell or squamous cell carcinoma (adequate wound healing is required prior to study entry)
    2. In situ carcinoma of the cervix or breast, treated curatively and without evidence of recurrence for at least 3 years prior to the study
    3. A primary malignancy which has been completely resected and in complete remission for ≥ 5 years
12. Simultaneously enrolled in any therapeutic clinical trial (except for long-term follow up studies)
13. Current or anticipating use of other anti-neoplastic or investigational agents while participating in this study
14. Either diagnosed with a psychiatric illness or under the impact of a social situation that would limit compliance with study requirements in the opinion of the investigator
15. Is pregnant or breastfeeding
16. Intolerance to the excipients of the cell product
17. Cardiac arrhythmia not controlled with medical management
18. Active COVID-19 (follow ASTCT guidelines)
19. Presence of active grade 2 to 4 acute, extensive chronic graft-versus-host disease (GVHD) or that require systemic steroids
20. Patients with active neurological auto immune or inflammatory disorders (e.g., Guillain-Barré Syndrome, Amyotrophic Lateral Sclerosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2040-03 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | Approximately 30 days
  The MTD is defined as the dose level immediately below that in which ≥ 2/6 participants experience a dose limiting toxicity (DLT).
Recommended Phase 2 Dose (RP2D) | Approximately 30 days
  Determine using MTD and DLTs.
Safety: Incidence of Serious Adverse Events/Adverse Events | Approximately 30 days
  Toxicities of DuoCAR20.19.22-D95 in combination with preceding lymphodepleting chemotherapy regimen As measured with CTCAE v 5.0,
Treatment-related Mortality (TRM) | Approximately 1 year
  defined by the absence of progressive disease at the time of death.
Presence of replication competent lentivirus (RCL) in peripheral blood samples | Approximately 15 years
  Measured with qPCR

SECONDARY OUTCOMES:
Efficacy of DuoCAR 20.19.22-D95 | up to 24 months
  Overall response rate defined by CR/PR rate as determined by WHO defined bone marrow results in ALL and the Lugano response criteria in B-cell NHL.
Safety related to DuoCAR20.19.22-D95 | Approximately 15 years
  To assess long-term safety risks, per FDA guidelines pertaining to gene therapy, as measured by delayed adverse events of special interest potentially related to DuoCAR20.19.22-D95
Pharmacology (Expansion kinetics) | 28 days
  Expansion kinetics of DuoCAR20.19.22-D95 over time as measured by PCR and/or flow cytometry, WinNonlin 8.4

CONTACTS AND LOCATIONS:
Overall Officials: Joseph McGuirk, D.O., Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Cancer Center, Westwood, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dioverti V, Boghdadly ZE, Shahid Z, Waghmare A, Abidi MZ, Pergam S, Boeckh M, Dadwal S, Kamboj M, Seo S, Chemaly RF, Papanicolaou GA. Revised Guidelines for Coronavirus Disease 19 Management in Hematopoietic Cell Transplantation and Cellular Therapy Recipients (August 2022). Transplant Cell Ther. 2022 Dec;28(12):810-821. doi: 10.1016/j.jtct.2022.09.002. Epub 2022 Sep 11. PMID 36103987
- [Background] Lee DW, Santomasso BD, Locke FL, Ghobadi A, Turtle CJ, Brudno JN, Maus MV, Park JH, Mead E, Pavletic S, Go WY, Eldjerou L, Gardner RA, Frey N, Curran KJ, Peggs K, Pasquini M, DiPersio JF, van den Brink MRM, Komanduri KV, Grupp SA, Neelapu SS. ASTCT Consensus Grading for Cytokine Release Syndrome and Neurologic Toxicity Associated with Immune Effector Cells. Biol Blood Marrow Transplant. 2019 Apr;25(4):625-638. doi: 10.1016/j.bbmt.2018.12.758. Epub 2018 Dec 25. PMID 30592986
- [Background] Wierda W, O'Brien S, Wen S, Faderl S, Garcia-Manero G, Thomas D, Do KA, Cortes J, Koller C, Beran M, Ferrajoli A, Giles F, Lerner S, Albitar M, Kantarjian H, Keating M. Chemoimmunotherapy with fludarabine, cyclophosphamide, and rituximab for relapsed and refractory chronic lymphocytic leukemia. J Clin Oncol. 2005 Jun 20;23(18):4070-8. doi: 10.1200/JCO.2005.12.516. Epub 2005 Mar 14. PMID 15767647
- [Background] Hedger MP, Meinhardt A. Local regulation of T cell numbers and lymphocyte-inhibiting activity in the interstitial tissue of the adult rat testis. J Reprod Immunol. 2000 Oct-Nov;48(2):69-80. doi: 10.1016/s0165-0378(00)00071-1. PMID 11011073
- [Background] Muller SM, Ege M, Pottharst A, Schulz AS, Schwarz K, Friedrich W. Transplacentally acquired maternal T lymphocytes in severe combined immunodeficiency: a study of 121 patients. Blood. 2001 Sep 15;98(6):1847-51. doi: 10.1182/blood.v98.6.1847. PMID 11535520
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Barrington SF, Mikhaeel NG, Kostakoglu L, Meignan M, Hutchings M, Mueller SP, Schwartz LH, Zucca E, Fisher RI, Trotman J, Hoekstra OS, Hicks RJ, O'Doherty MJ, Hustinx R, Biggi A, Cheson BD. Role of imaging in the staging and response assessment of lymphoma: consensus of the International Conference on Malignant Lymphomas Imaging Working Group. J Clin Oncol. 2014 Sep 20;32(27):3048-58. doi: 10.1200/JCO.2013.53.5229. PMID 25113771
- [Background] Pulsipher MA, Han X, Maude SL, Laetsch TW, Qayed M, Rives S, Boyer MW, Hiramatsu H, Yanik GA, Driscoll T, Myers GD, Bader P, Baruchel A, Buechner J, Stefanski HE, Kalfoglou C, Nguyen K, Waldron ER, Thudium Mueller K, Maier HJ, Kari G, Grupp SA. Next-Generation Sequencing of Minimal Residual Disease for Predicting Relapse after Tisagenlecleucel in Children and Young Adults with Acute Lymphoblastic Leukemia. Blood Cancer Discov. 2022 Jan;3(1):66-81. doi: 10.1158/2643-3230.BCD-21-0095. Epub 2021 Dec 1. PMID 35019853
- [Background] Rossoff J, Baggott C, Prabhu S, Pacenta H, Phillips CL, Stefanski H, Talano JA, Moskop A, Margossian SP, Verneris MR, Myers GD, Karras N, Brown PA, Qayed M, Hermiston M, Satwani P, Krupski C, Keating AK, Wilcox R, Rabik CA, Fabrizio VA, Kunicki M, Chinnabhandar V, Goksenin AY, Curran KJ, Mackall CL, Laetsch TW, Schultz LM. Out-of-specification tisagenlecleucel does not compromise safety or efficacy in pediatric acute lymphoblastic leukemia. Blood. 2021 Nov 25;138(21):2138-2142. doi: 10.1182/blood.2021012392. No abstract available. PMID 34499715
- [Background] Laetsch TW, Myers GD, Baruchel A, Dietz AC, Pulsipher MA, Bittencourt H, Buechner J, De Moerloose B, Davis KL, Nemecek E, Driscoll T, Mechinaud F, Boissel N, Rives S, Bader P, Peters C, Sabnis HS, Grupp SA, Yanik GA, Hiramatsu H, Stefanski HE, Rasouliyan L, Yi L, Shah S, Zhang J, Harris AC. Patient-reported quality of life after tisagenlecleucel infusion in children and young adults with relapsed or refractory B-cell acute lymphoblastic leukaemia: a global, single-arm, phase 2 trial. Lancet Oncol. 2019 Dec;20(12):1710-1718. doi: 10.1016/S1470-2045(19)30493-0. Epub 2019 Oct 9. PMID 31606419
- [Background] Gardner RA, Finney O, Annesley C, Brakke H, Summers C, Leger K, Bleakley M, Brown C, Mgebroff S, Kelly-Spratt KS, Hoglund V, Lindgren C, Oron AP, Li D, Riddell SR, Park JR, Jensen MC. Intent-to-treat leukemia remission by CD19 CAR T cells of defined formulation and dose in children and young adults. Blood. 2017 Jun 22;129(25):3322-3331. doi: 10.1182/blood-2017-02-769208. Epub 2017 Apr 13. PMID 28408462
- [Background] Schneider D, Xiong Y, Wu D, Hu P, Alabanza L, Steimle B, Mahmud H, Anthony-Gonda K, Krueger W, Zhu Z, Dimitrov DS, Orentas RJ, Dropulic B. Trispecific CD19-CD20-CD22-targeting duoCAR-T cells eliminate antigen-heterogeneous B cell tumors in preclinical models. Sci Transl Med. 2021 Mar 24;13(586):eabc6401. doi: 10.1126/scitranslmed.abc6401. PMID 33762438
- [Background] Dekker L, Calkoen FG, Jiang Y, Blok H, Veldkamp SR, De Koning C, Spoon M, Admiraal R, Hoogerbrugge P, Vormoor B, Vormoor HJ, Visscher H, Bierings M, Van Der Vlugt M, Van Tinteren H, Nijstad AL, Huitema ADR, Van Der Elst KCM, Pieters R, Lindemans CA, Nierkens S. Fludarabine exposure predicts outcome after CD19 CAR T-cell therapy in children and young adults with acute leukemia. Blood Adv. 2022 Apr 12;6(7):1969-1976. doi: 10.1182/bloodadvances.2021006700. PMID 35134115
- [Background] Rogers PR, Song J, Gramaglia I, Killeen N, Croft M. OX40 promotes Bcl-xL and Bcl-2 expression and is essential for long-term survival of CD4 T cells. Immunity. 2001 Sep;15(3):445-55. doi: 10.1016/s1074-7613(01)00191-1. PMID 11567634
- [Background] Gramaglia I, Jember A, Pippig SD, Weinberg AD, Killeen N, Croft M. The OX40 costimulatory receptor determines the development of CD4 memory by regulating primary clonal expansion. J Immunol. 2000 Sep 15;165(6):3043-50. doi: 10.4049/jimmunol.165.6.3043. PMID 10975814
- [Background] Maxwell JR, Weinberg A, Prell RA, Vella AT. Danger and OX40 receptor signaling synergize to enhance memory T cell survival by inhibiting peripheral deletion. J Immunol. 2000 Jan 1;164(1):107-12. doi: 10.4049/jimmunol.164.1.107. PMID 10605000
- [Background] Rafiq S, Hackett CS, Brentjens RJ. Engineering strategies to overcome the current roadblocks in CAR T cell therapy. Nat Rev Clin Oncol. 2020 Mar;17(3):147-167. doi: 10.1038/s41571-019-0297-y. Epub 2019 Dec 17. PMID 31848460
- [Background] Pasquini MC, Hu ZH, Curran K, Laetsch T, Locke F, Rouce R, Pulsipher MA, Phillips CL, Keating A, Frigault MJ, Salzberg D, Jaglowski S, Sasine JP, Rosenthal J, Ghosh M, Landsburg D, Margossian S, Martin PL, Kamdar MK, Hematti P, Nikiforow S, Turtle C, Perales MA, Steinert P, Horowitz MM, Moskop A, Pacaud L, Yi L, Chawla R, Bleickardt E, Grupp S. Real-world evidence of tisagenlecleucel for pediatric acute lymphoblastic leukemia and non-Hodgkin lymphoma. Blood Adv. 2020 Nov 10;4(21):5414-5424. doi: 10.1182/bloodadvances.2020003092. PMID 33147337
- [Background] Frigault MJ, Maus MV. State of the art in CAR T cell therapy for CD19+ B cell malignancies. J Clin Invest. 2020 Apr 1;130(4):1586-1594. doi: 10.1172/JCI129208. PMID 32235098
- [Background] Moreno-Cortes E, Franco-Fuquen P, Garcia-Robledo JE, Forero J, Booth N, Castro JE. ICOS and OX40 tandem co-stimulation enhances CAR T-cell cytotoxicity and promotes T-cell persistence phenotype. Front Oncol. 2023 Aug 18;13:1200914. doi: 10.3389/fonc.2023.1200914. eCollection 2023. PMID 37719008
- [Background] Fabrizio VA, Boelens JJ, Mauguen A, Baggott C, Prabhu S, Egeler E, Mavroukakis S, Pacenta H, Phillips CL, Rossoff J, Stefanski HE, Talano JA, Moskop A, Margossian SP, Verneris MR, Myers GD, Karras NA, Brown PA, Qayed M, Hermiston M, Satwani P, Krupski C, Keating AK, Wilcox R, Rabik CA, Chinnabhandar V, Kunicki M, Goksenin AY, Mackall CL, Laetsch TW, Schultz LM, Curran KJ. Optimal fludarabine lymphodepletion is associated with improved outcomes after CAR T-cell therapy. Blood Adv. 2022 Apr 12;6(7):1961-1968. doi: 10.1182/bloodadvances.2021006418. PMID 34788386
- [Background] Hines MR, Knight TE, McNerney KO, Leick MB, Jain T, Ahmed S, Frigault MJ, Hill JA, Jain MD, Johnson WT, Lin Y, Mahadeo KM, Maron GM, Marsh RA, Neelapu SS, Nikiforow S, Ombrello AK, Shah NN, Talleur AC, Turicek D, Vatsayan A, Wong SW, Maus MV, Komanduri KV, Berliner N, Henter JI, Perales MA, Frey NV, Teachey DT, Frank MJ, Shah NN. Immune Effector Cell-Associated Hemophagocytic Lymphohistiocytosis-Like Syndrome. Transplant Cell Ther. 2023 Jul;29(7):438.e1-438.e16. doi: 10.1016/j.jtct.2023.03.006. Epub 2023 Mar 9. PMID 36906275
- [Background] Poe JC, Minard-Colin V, Kountikov EI, Haas KM, Tedder TF. A c-Myc and surface CD19 signaling amplification loop promotes B cell lymphoma development and progression in mice. J Immunol. 2012 Sep 1;189(5):2318-25. doi: 10.4049/jimmunol.1201000. Epub 2012 Jul 23. PMID 22826319
- [Background] Fruman DA. Phosphoinositide 3-kinase and its targets in B-cell and T-cell signaling. Curr Opin Immunol. 2004 Jun;16(3):314-20. doi: 10.1016/j.coi.2004.03.014. PMID 15134780
- [Background] Rogel A, Willoughby JE, Buchan SL, Leonard HJ, Thirdborough SM, Al-Shamkhani A. Akt signaling is critical for memory CD8+ T-cell development and tumor immune surveillance. Proc Natl Acad Sci U S A. 2017 Feb 14;114(7):E1178-E1187. doi: 10.1073/pnas.1611299114. Epub 2017 Jan 30. PMID 28137869
- [Background] Gravestein LA, Nieland JD, Kruisbeek AM, Borst J. Novel mAbs reveal potent co-stimulatory activity of murine CD27. Int Immunol. 1995 Apr;7(4):551-7. doi: 10.1093/intimm/7.4.551. PMID 7547681
- [Background] Liakou CI, Kamat A, Tang DN, Chen H, Sun J, Troncoso P, Logothetis C, Sharma P. CTLA-4 blockade increases IFNgamma-producing CD4+ICOShi cells to shift the ratio of effector to regulatory T cells in cancer patients. Proc Natl Acad Sci U S A. 2008 Sep 30;105(39):14987-92. doi: 10.1073/pnas.0806075105. Epub 2008 Sep 25. PMID 18818309
- [Background] Haas KM, Sen S, Sanford IG, Miller AS, Poe JC, Tedder TF. CD22 ligand binding regulates normal and malignant B lymphocyte survival in vivo. J Immunol. 2006 Sep 1;177(5):3063-73. doi: 10.4049/jimmunol.177.5.3063. PMID 16920943
- [Background] Hombach AA, Heiders J, Foppe M, Chmielewski M, Abken H. OX40 costimulation by a chimeric antigen receptor abrogates CD28 and IL-2 induced IL-10 secretion by redirected CD4(+) T cells. Oncoimmunology. 2012 Jul 1;1(4):458-466. doi: 10.4161/onci.19855. PMID 22754764
- [Background] Majzner RG, Mackall CL. Tumor Antigen Escape from CAR T-cell Therapy. Cancer Discov. 2018 Oct;8(10):1219-1226. doi: 10.1158/2159-8290.CD-18-0442. Epub 2018 Aug 22. PMID 30135176
- [Background] Shah NN, Maatman T, Hari P, Johnson B. Multi Targeted CAR-T Cell Therapies for B-Cell Malignancies. Front Oncol. 2019 Mar 12;9:146. doi: 10.3389/fonc.2019.00146. eCollection 2019. PMID 30915277
- [Background] Holland EM, Molina JC, Dede K, Moyer D, Zhou T, Yuan CM, Wang HW, Stetler-Stevenson M, Mackall C, Fry TJ, Panch S, Highfill S, Stroncek D, Little L, Lee DW, Shalabi H, Yates B, Shah N. Efficacy of second CAR-T (CART2) infusion limited by poor CART expansion and antigen modulation. J Immunother Cancer. 2022 May;10(5):e004483. doi: 10.1136/jitc-2021-004483. PMID 35534047
- [Background] Cao Y, Xiao Y, Wang N, Wang G, Huang L, Hong Z, Meng L, Zhou X, Wang J, Yang Y, Xu H, Zhang S, Xiao M, Chen L, Zheng M, Li C, Mao X, Gu C, Zhang T, Zhang Y, Zhou J. CD19/CD22 Chimeric Antigen Receptor T Cell Cocktail Therapy following Autologous Transplantation in Patients with Relapsed/Refractory Aggressive B Cell Lymphomas. Transplant Cell Ther. 2021 Nov;27(11):910.e1-910.e11. doi: 10.1016/j.jtct.2021.08.012. Epub 2021 Aug 20. PMID 34425260
- [Background] Fry TJ, Shah NN, Orentas RJ, Stetler-Stevenson M, Yuan CM, Ramakrishna S, Wolters P, Martin S, Delbrook C, Yates B, Shalabi H, Fountaine TJ, Shern JF, Majzner RG, Stroncek DF, Sabatino M, Feng Y, Dimitrov DS, Zhang L, Nguyen S, Qin H, Dropulic B, Lee DW, Mackall CL. CD22-targeted CAR T cells induce remission in B-ALL that is naive or resistant to CD19-targeted CAR immunotherapy. Nat Med. 2018 Jan;24(1):20-28. doi: 10.1038/nm.4441. Epub 2017 Nov 20. PMID 29155426
- [Background] Pan J, Niu Q, Deng B, Liu S, Wu T, Gao Z, Liu Z, Zhang Y, Qu X, Zhang Y, Liu S, Ling Z, Lin Y, Zhao Y, Song Y, Tan X, Zhang Y, Li Z, Yin Z, Chen B, Yu X, Yan J, Zheng Q, Zhou X, Gao J, Chang AH, Feng X, Tong C. CD22 CAR T-cell therapy in refractory or relapsed B acute lymphoblastic leukemia. Leukemia. 2019 Dec;33(12):2854-2866. doi: 10.1038/s41375-019-0488-7. Epub 2019 May 20. PMID 31110217
- [Background] Locke FL, Ghobadi A, Jacobson CA, Miklos DB, Lekakis LJ, Oluwole OO, Lin Y, Braunschweig I, Hill BT, Timmerman JM, Deol A, Reagan PM, Stiff P, Flinn IW, Farooq U, Goy A, McSweeney PA, Munoz J, Siddiqi T, Chavez JC, Herrera AF, Bartlett NL, Wiezorek JS, Navale L, Xue A, Jiang Y, Bot A, Rossi JM, Kim JJ, Go WY, Neelapu SS. Long-term safety and activity of axicabtagene ciloleucel in refractory large B-cell lymphoma (ZUMA-1): a single-arm, multicentre, phase 1-2 trial. Lancet Oncol. 2019 Jan;20(1):31-42. doi: 10.1016/S1470-2045(18)30864-7. Epub 2018 Dec 2. PMID 30518502
- [Background] Fayad L, Offner F, Smith MR, Verhoef G, Johnson P, Kaufman JL, Rohatiner A, Advani A, Foran J, Hess G, Coiffier B, Czuczman M, Gine E, Durrant S, Kneissl M, Luu KT, Hua SY, Boni J, Vandendries E, Dang NH. Safety and clinical activity of a combination therapy comprising two antibody-based targeting agents for the treatment of non-Hodgkin lymphoma: results of a phase I/II study evaluating the immunoconjugate inotuzumab ozogamicin with rituximab. J Clin Oncol. 2013 Feb 10;31(5):573-83. doi: 10.1200/JCO.2012.42.7211. Epub 2013 Jan 7. PMID 23295790
- [Background] Rigaud C, Auperin A, Jourdain A, Haouy S, Couec ML, Aladjidi N, Gandemer V, Lambliotte A, Plat G, Landman-Parker J, Michon J, Leblanc T, Patte C, Minard-Colin V. Outcome of relapse in children and adolescents with B-cell non-Hodgkin lymphoma and mature acute leukemia: A report from the French LMB study. Pediatr Blood Cancer. 2019 Sep;66(9):e27873. doi: 10.1002/pbc.27873. Epub 2019 Jun 17. PMID 31207026
- [Background] Hochberg J, El-Mallawany NK, Abla O. Adolescent and young adult non-Hodgkin lymphoma. Br J Haematol. 2016 May;173(4):637-50. doi: 10.1111/bjh.14074. Epub 2016 Apr 12. PMID 27071675
- [Background] Anoop P, Sankpal S, Stiller C, Tewari S, Lancaster DL, Khabra K, Taj MM. Outcome of childhood relapsed or refractory mature B-cell non-Hodgkin lymphoma and acute lymphoblastic leukemia. Leuk Lymphoma. 2012 Oct;53(10):1882-8. doi: 10.3109/10428194.2012.677534. Epub 2012 Apr 23. PMID 22448922
- [Background] Egan G, Goldman S, Alexander S. Mature B-NHL in children, adolescents and young adults: current therapeutic approach and emerging treatment strategies. Br J Haematol. 2019 Jun;185(6):1071-1085. doi: 10.1111/bjh.15734. Epub 2019 Jan 6. PMID 30613948
- [Background] Cairo M, Auperin A, Perkins SL, Pinkerton R, Harrison L, Goldman S, Patte C. Overall survival of children and adolescents with mature B cell non-Hodgkin lymphoma who had refractory or relapsed disease during or after treatment with FAB/LMB 96: A report from the FAB/LMB 96 study group. Br J Haematol. 2018 Sep;182(6):859-869. doi: 10.1111/bjh.15491. Epub 2018 Jul 9. PMID 29984828
- [Background] Moleti ML, Testi AM, Foa R. Treatment of relapsed/refractory paediatric aggressive B-cell non-Hodgkin lymphoma. Br J Haematol. 2020 Jun;189(5):826-843. doi: 10.1111/bjh.16461. Epub 2020 Mar 6. PMID 32141616
- [Background] Rytting ME, Thomas DA, O'Brien SM, Ravandi-Kashani F, Jabbour EJ, Franklin AR, Kadia TM, Pemmaraju N, Daver NG, Ferrajoli A, Garcia-Manero G, Konopleva MY, Cortes JE, Borthakur G, Garris R, Cardenas-Turanzas M, Schroeder K, Jorgensen JL, Kornblau SM, Kantarjian HM. Augmented Berlin-Frankfurt-Munster therapy in adolescents and young adults (AYAs) with acute lymphoblastic leukemia (ALL). Cancer. 2014 Dec 1;120(23):3660-8. doi: 10.1002/cncr.28930. Epub 2014 Jul 17. PMID 25042398
- [Background] Ram R, Wolach O, Vidal L, Gafter-Gvili A, Shpilberg O, Raanani P. Adolescents and young adults with acute lymphoblastic leukemia have a better outcome when treated with pediatric-inspired regimens: systematic review and meta-analysis. Am J Hematol. 2012 May;87(5):472-8. doi: 10.1002/ajh.23149. Epub 2012 Mar 3. PMID 22388572
- [Background] Essig S, Li Q, Chen Y, Hitzler J, Leisenring W, Greenberg M, Sklar C, Hudson MM, Armstrong GT, Krull KR, Neglia JP, Oeffinger KC, Robison LL, Kuehni CE, Yasui Y, Nathan PC. Risk of late effects of treatment in children newly diagnosed with standard-risk acute lymphoblastic leukaemia: a report from the Childhood Cancer Survivor Study cohort. Lancet Oncol. 2014 Jul;15(8):841-51. doi: 10.1016/S1470-2045(14)70265-7. Epub 2014 Jun 19. PMID 24954778
- [Background] Hunger SP, Baruchel A, Biondi A, Evans WE, Jeha S, Loh M, Moericke A, Pieters R, Relling MV, Schmiegelow K, Schrappe M, Silverman LB, Stanulla M, Valsecchi MG, Vora A, Pui CH. The thirteenth international childhood acute lymphoblastic leukemia workshop report: La Jolla, CA, USA, December 7-9, 2011. Pediatr Blood Cancer. 2013 Feb;60(2):344-8. doi: 10.1002/pbc.24354. Epub 2012 Sep 28. No abstract available. PMID 23024117
- [Background] Faderl S, O'Brien S, Pui CH, Stock W, Wetzler M, Hoelzer D, Kantarjian HM. Adult acute lymphoblastic leukemia: concepts and strategies. Cancer. 2010 Mar 1;116(5):1165-76. doi: 10.1002/cncr.24862. PMID 20101737
- [Background] Cheson BD, Fisher RI, Barrington SF, Cavalli F, Schwartz LH, Zucca E, Lister TA; Alliance, Australasian Leukaemia and Lymphoma Group; Eastern Cooperative Oncology Group; European Mantle Cell Lymphoma Consortium; Italian Lymphoma Foundation; European Organisation for Research; Treatment of Cancer/Dutch Hemato-Oncology Group; Grupo Espanol de Medula Osea; German High-Grade Lymphoma Study Group; German Hodgkin's Study Group; Japanese Lymphorra Study Group; Lymphoma Study Association; NCIC Clinical Trials Group; Nordic Lymphoma Study Group; Southwest Oncology Group; United Kingdom National Cancer Research Institute. Recommendations for initial evaluation, staging, and response assessment of Hodgkin and non-Hodgkin lymphoma: the Lugano classification. J Clin Oncol. 2014 Sep 20;32(27):3059-68. doi: 10.1200/JCO.2013.54.8800. PMID 25113753
- [Background] Gill S, Carney D, Ritchie D, Wolf M, Westerman D, Prince HM, Januszewicz H, Seymour JF. The frequency, manifestations, and duration of prolonged cytopenias after first-line fludarabine combination chemotherapy. Ann Oncol. 2010 Feb;21(2):331-334. doi: 10.1093/annonc/mdp297. Epub 2009 Jul 22. PMID 19625344
- [Background] Fried S, Avigdor A, Bielorai B, Meir A, Besser MJ, Schachter J, Shimoni A, Nagler A, Toren A, Jacoby E. Early and late hematologic toxicity following CD19 CAR-T cells. Bone Marrow Transplant. 2019 Oct;54(10):1643-1650. doi: 10.1038/s41409-019-0487-3. Epub 2019 Feb 26. PMID 30809033
- [Background] Levine JE, Grupp SA, Pulsipher MA, Dietz AC, Rives S, Myers GD, August KJ, Verneris MR, Buechner J, Laetsch TW, Bittencourt H, Baruchel A, Boyer MW, De Moerloose B, Qayed M, Davies SM, Phillips CL, Driscoll TA, Bader P, Schlis K, Wood PA, Mody R, Yi L, Leung M, Eldjerou LK, June CH, Maude SL. Pooled safety analysis of tisagenlecleucel in children and young adults with B cell acute lymphoblastic leukemia. J Immunother Cancer. 2021 Aug;9(8):e002287. doi: 10.1136/jitc-2020-002287. PMID 34353848
- [Background] Schuster, SJ, Svoboda J, Nasta SD, et al, Sustained Remissions Following Chimeric Antigen Receptor Modified T Cells Directed Against CD19 (CTL019) in Patients with Relapsed or Refractory CD19+ Lymphomas. Blood, 2015. 126(23): p. 183-183.
- [Background] Jourdain A, Auperin A, Minard-Colin V, Aladjidi N, Zsiros J, Coze C, Gandemer V, Bertrand Y, Leverger G, Bergeron C, Michon J, Patte C; SFCE LNH Committee. Outcome of and prognostic factors for relapse in children and adolescents with mature B-cell lymphoma and leukemia treated in three consecutive prospective "Lymphomes Malins B" protocols. A Societe Francaise des Cancers de l'Enfant study. Haematologica. 2015 Jun;100(6):810-7. doi: 10.3324/haematol.2014.121434. Epub 2015 Feb 27. PMID 25724577
- [Background] Guedan S, Chen X, Madar A, Carpenito C, McGettigan SE, Frigault MJ, Lee J, Posey AD Jr, Scholler J, Scholler N, Bonneau R, June CH. ICOS-based chimeric antigen receptors program bipolar TH17/TH1 cells. Blood. 2014 Aug 14;124(7):1070-80. doi: 10.1182/blood-2013-10-535245. Epub 2014 Jul 1. PMID 24986688
- [Background] Porter DL, Hwang WT, Frey NV, Lacey SF, Shaw PA, Loren AW, Bagg A, Marcucci KT, Shen A, Gonzalez V, Ambrose D, Grupp SA, Chew A, Zheng Z, Milone MC, Levine BL, Melenhorst JJ, June CH. Chimeric antigen receptor T cells persist and induce sustained remissions in relapsed refractory chronic lymphocytic leukemia. Sci Transl Med. 2015 Sep 2;7(303):303ra139. doi: 10.1126/scitranslmed.aac5415. PMID 26333935
- [Background] Kawalekar OU, O'Connor RS, Fraietta JA, Guo L, McGettigan SE, Posey AD Jr, Patel PR, Guedan S, Scholler J, Keith B, Snyder NW, Blair IA, Milone MC, June CH. Distinct Signaling of Coreceptors Regulates Specific Metabolism Pathways and Impacts Memory Development in CAR T Cells. Immunity. 2016 Feb 16;44(2):380-90. doi: 10.1016/j.immuni.2016.01.021. PMID 26885860
- [Background] Zhao Z, Condomines M, van der Stegen SJC, Perna F, Kloss CC, Gunset G, Plotkin J, Sadelain M. Structural Design of Engineered Costimulation Determines Tumor Rejection Kinetics and Persistence of CAR T Cells. Cancer Cell. 2015 Oct 12;28(4):415-428. doi: 10.1016/j.ccell.2015.09.004. PMID 26461090
- [Background] Long AH, Haso WM, Shern JF, Wanhainen KM, Murgai M, Ingaramo M, Smith JP, Walker AJ, Kohler ME, Venkateshwara VR, Kaplan RN, Patterson GH, Fry TJ, Orentas RJ, Mackall CL. 4-1BB costimulation ameliorates T cell exhaustion induced by tonic signaling of chimeric antigen receptors. Nat Med. 2015 Jun;21(6):581-90. doi: 10.1038/nm.3838. Epub 2015 May 4. PMID 25939063
- [Background] Turtle CJ, Hanafi LA, Berger C, Gooley TA, Cherian S, Hudecek M, Sommermeyer D, Melville K, Pender B, Budiarto TM, Robinson E, Steevens NN, Chaney C, Soma L, Chen X, Yeung C, Wood B, Li D, Cao J, Heimfeld S, Jensen MC, Riddell SR, Maloney DG. CD19 CAR-T cells of defined CD4+:CD8+ composition in adult B cell ALL patients. J Clin Invest. 2016 Jun 1;126(6):2123-38. doi: 10.1172/JCI85309. Epub 2016 Apr 25. PMID 27111235
- [Background] Lee DW, Kochenderfer JN, Stetler-Stevenson M, Cui YK, Delbrook C, Feldman SA, Fry TJ, Orentas R, Sabatino M, Shah NN, Steinberg SM, Stroncek D, Tschernia N, Yuan C, Zhang H, Zhang L, Rosenberg SA, Wayne AS, Mackall CL. T cells expressing CD19 chimeric antigen receptors for acute lymphoblastic leukaemia in children and young adults: a phase 1 dose-escalation trial. Lancet. 2015 Feb 7;385(9967):517-528. doi: 10.1016/S0140-6736(14)61403-3. Epub 2014 Oct 13. PMID 25319501
- [Background] National Institute of Health/National Cancer Institute - Cancer Therapy Evaluation Program (CTEP). Common Terminology Criteria for Adverse Events (CTCAE). URL: https://ctep.cancer.gov/protocoldevelopment/electronic_applications/ctc.htm#ctc_60 Accessed 01-26-2022